CLINICAL TRIAL: NCT00275249
Title: Evolution of Analgesic Tolerance During Long Term Treatment of Chronic Pain With Opioids
Brief Title: Evolution of Analgesic Tolerance With Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: H5612-23841
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Pain
Keywords: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Levorphanol

INTERVENTIONS:
Drug: levorphanol

SUMMARY:
The purpose of this study is to determine the extent to which analgesic tolerance develops in chronic pain patients who are either started on opioids or who receive an increase in pre-study opioid dose level and then observed during long-term (20 weeks) stable opioid therapy. In addition to clinical measures of relief of ongoing chronic pain, estimation of tolerance development will be supplemented by periodic assessment of the anti-nociceptive effects of opioids using the brief thermal sensitization model.

DETAILED DESCRIPTION:
The purpose of this study is to determine the extent to which analgesic tolerance develops in chronic pain patients who are either started on opioids or who receive an increase in pre-study opioid dose level and then observed during long-term (20 weeks) stable opioid therapy. In addition to clinical measures of relief of ongoing chronic pain, estimation of tolerance development will be supplemented by periodic assessment of the anti-nociceptive effects of opioids using the brief thermal sensitization model.

ELIGIBILITY:
Inclusion Criteria:

1. Adults who are 21-80 years of age.
2. Desires opioid dose increase (with approval of current prescribing physician), or is not on opioids and desires a trial of opioids for ongoing pain.
3. Expected to remain in stable health for at least a six months period surrounding study participation.
4. Able and willing to provide written informed consent.
5. Able to understand and follow the instructions of the investigator, including all rating scales.
6. Stable chronic pain that is either neuropathic or non-neuropathic in origin as defined above. The diagnosis will be based on history, physical examination, and review of medical records confirming the diagnosis.
7. For a chronic user: stable opioid use of between 31 and 150 mg/day morphine equivalent. Stable use is defined as no change in the daily dose of opioids for the month preceding study entry.
8. For naïve users: have not used opioids or use is less than or equal to 30 mg/day morphine equivalent for their chronic pain.
9. Chronic pain must be at least moderately severe, defined as an average daily pain severity exceeding 40 mm on a 100 mm pain intensity visual analog scale (VAS).
10. Female subjects must be post-menopausal, physically incapable of becoming pregnant, or using acceptable birth control method. Acceptable methods of birth control include hormonal contraceptives or double-barrier methods (condom or diaphragm with spermicidal agent or IUD). If practicing an acceptable method of birth control, confirmation of negative pregnancy urine test for female subjects is required at the Screening Visit. No special precautions are required for male subjects because levorphanol is an approved therapy for chronic pain.

Exclusion Criteria:

1. Use of opioid mixed agonist-antagonists (pentazocine, buprenorphine, butorphanol), or tramadol, will not be allowed. Use of an intrathecal opioid infusion pump will not be allowed.
2. Allergy to levorphanol.
3. Patients who are unable to read or speak English.
4. A pain complaint, which is believed to be psychogenic in nature or cannot be confirmed by medical records and physical examination.
5. Pain due to a disease, such as cancer not in remission, which is expected to substantially progress during the study period.
6. Cognitive impairment, psychiatric disorder, or unrelated neurological disorder severe enough to interfere with assessment of pain and sensory systems.
7. Pregnancy.
8. Has received an investigational drug within 30 days prior to Study Visit 2.
9. A current substance abuse disorder, a positive urine drug screen, or a history of opioid drug abuse at any time in the past.
10. Intolerable side effects, or failed to achieve adequate analgesic effect during prior attempts at opioid dose escalation within the range of doses to be used in this study.
11. Co-existing medical conditions or required medication use that contraindicate study procedures or opioid dose escalation. Subjects with disorders, such as unusual skin fragility or severe peripheral neuropathy that contraindicate brief thermal sensitization will be allowed to participate without this component.
12. Those, in the opinion of the investigator, who are unlikely to comply with the study protocol or who are unsuitable for any other reason.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-03; Primary Completion 2004-10 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rowbotham, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Pain Clinical Research Center, San Francisco, California, United States

REFERENCES:
- [Derived] Rowbotham MC, Wallace M. Evolution of Analgesic Tolerance and Opioid-Induced Hyperalgesia Over 6 Months: Double-Blind Randomized Trial Incorporating Experimental Pain Models. J Pain. 2020 Sep-Oct;21(9-10):1031-1046. doi: 10.1016/j.jpain.2020.01.005. Epub 2020 Feb 1. PMID 32006699